CLINICAL TRIAL: NCT03657836
Title: Evaluation of Effectiveness of the Sublimated Mare Milk Supplement in Protection of Gut Mucosal Lining During Antibiotic Treatment
Brief Title: The Sublimated Mare Milk Supplement's Effect on Gut Mucosal Lining After Antibiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nazarbayev University Medical Center (Other)
Collaborators: Eurasia Invest Ltd. (Industry); Ministry of Education and Science, Republic of Kazakhstan (Other Government)
Responsible Party: Principal Investigator, Almagul Kushugulova, Head of the Laboratory of Human Microbiome and Longevity, Nazarbayev University Medical Center
Organization: Nazarbayev University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP05135073
Record Dates: First submitted 2018-08-29; First posted 2018-09-05 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Acute Bronchitis
Keywords: Acute Bronchitis; Mare milk; Gut mucosa; Antibiotics
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement and antibiotics (Experimental): Participants will take a supplement of 1 sachet (20 mg) dissolved in 200 ml of warm water (36-37 °C) once a day for 60 days accompanied with the standard antibiotic therapy (cefuroxime and ceftriaxone) up to 7 days.
  Interventions: Dietary Supplement: Sublimated mare milk supplement; Drug: Standard antibiotic therapy
- Antibiotics only (Other): Participants will take the prescribed antibiotic therapy (cefuroxime and ceftriaxone) up to 7 days.
  Interventions: Drug: Standard antibiotic therapy

INTERVENTIONS:
Dietary Supplement: Sublimated mare milk supplement — The dietary supplement consisting of sublimated mare milk packed in single-dose sachet.
  Arms: Dietary supplement and antibiotics
Drug: Standard antibiotic therapy — Patients will be given standard therapy antibiotics cefuroxime and ceftriaxone for up to 7 days period.

SUMMARY:
This clinical trial studies the effect of sublimated mare milk supplement on gut microbiome of patients with acute bronchitis.

DETAILED DESCRIPTION:
Food has a significant effect on the health of the body, the relationship between diet and health actualizes the importance of expanding the research of functional products. In mare's milk contains about 40 biological components necessary for the human body: amino acids, fats, enzymes (lysozyme, amylase), microelements (calcium, sodium, potassium, phosphorus, iron, magnesium, copper, iodine, sulfur, cobalt, zinc, bromine) and vitamins (A, C, B1, B2, B6, B12, E, H, PP, beta-carotene, folic acid) in optimally balanced proportions.

A high percentage of nutrients, including vitamins, amino acids, contribute to immunomodulation, increasing the adaptogenic properties of the body. Valiev A demonstrated the effect of the essential fatty acids of mare's milk on immunocompetent cells and non-specific resistance after 6 weeks from the beginning of inclusion in the ration of mare's milk.

Secretory IgA is the main immunoglobulin of mare's milk. The homology of human secretory IgA and mare's was previously demonstrated by cross-reactions using human anti-IgA antiserum.

The mare's milk has a powerful detoxification effect, the mare's microflora neutralizes the effect of mutagens, possesses, replenishes with the necessary complex of nutrients and removes toxins from the body. The milk has a certain degree of antimicrobial effect in relation to opportunistic and pathogenic fungi, bacteria and viruses due to its own microflora.

The mare's milk is rich in active substances, natural enzymes that help regulate intestinal flora, limiting the growth of unwanted bacteria and increasing the growth of bifidobacteria and lactic acid bacteria.

In addition, the composition of mare's milk provided immunoglobulins A, M and G, which act as a marker of those microorganisms that can be pathogenic, which facilitates the protection task.

The high antimicrobial activity of mare's milk is associated with the lysozyme contained in it, immunoglobulins, lactoperoxidase and lactoferrin. Getting into the digestive tract lysozyme has a powerful normalizing effect on the composition of the microbial flora of the mouth and intestines. Lysozyme of breast milk is 100 times more active than lysozyme of cow's milk. It not only inhibits the growth of pathogenic flora, but also promotes the growth of bifidoflora in the intestines of infants.

In the framework of the project, methods for the restoration of the mucos layer of the intestine after antibiotic therapy will be developed. In order to develop the algorithm, preliminary studies will be made of changes in the structure of the intestinal microbiota after antibiotic therapy. Recruiting of patients with infectious / non-infectious pathology is supposed, clinical and laboratory examination, biomaterial sampling during antibiotic therapy, 1-5 days and 1-60 days after completion will be performed. Along with the study of microflora, local immunity studies will be carried out. To study the fundamental foundations, experimental studies will be carried out on laboratory animals. On the basis of the knowledge obtained, an algorithm for the restoration of the mucinous layer of the intestine after antibiotic therapy will be published in the form of methodological recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged 4-5 years
* The voluntary informed consent of the parent to participate in the study
* Established diagnosis of acute upper respiratory tract disease with prescription of antibacterial therapy
* The duration of symptoms of acute upper respiratory tract disease no more than 72 hours
* Lack of prescription of antibacterial drugs in the last 3 months

Exclusion Criteria:

* Severe forms of acute infections
* The presence in the history of taking probiotics and antibiotics for three months before admission to hospital
* Presence in the anamnesis of chronic diseases of the digestive tract, and also of any surgeries on the digestive tract
* The presence of severe concomitant diseases of the kidneys, liver, cardiovascular, respiratory and other body systems, cancer, mental and decompensated endocrine diseases, tuberculosis, HIV infection
* Patient involvement in other clinical trials within the last 3 months
* Lack of willingness of the patient to cooperate with the doctor-researcher

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in intestinal microbial composition | Baseline, Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 10, Day 15, Day 20, Day 25, Day 30, Day 35, Day 40, Day 45, Day 50, Day 55, Day 60
  Rectal swabs will be taken for further analysis of DNA sequence with MiSeq Reporter PCR Amplicon.
Changes in intestinal immune status biomarkers. | Baseline, Day 60
  Levels of immune markers (cytokines, secretory Immunoglobulin A, interleukins) will be assessed from stool samples.

SECONDARY OUTCOMES:
Changes in weight of the patient | Baseline, Day 60
  Weight will be assessed according to percentile tables
Defecation frequency | Baseline, up to 60 days
  Defecation frequency based on patient's/parent's/guardian's reports over period of 60 days
Changes in consistency of stool | Baseline, Day 60
  Consistency of stool will be evaluated according to Bristol scale with severe hard lumps and liquid stool being a severe constipation (Type 1) and severe diarrhea (Type 7) respectively.
Changes in color of stool, | Baseline, Day 60
  Stool color changes will be assessed based on baseline and final visit (Day 60).

CONTACTS AND LOCATIONS:
Overall Officials: Almagul Kushugulova, MD, PhD, Principal Investigator — National Laboratory Astana
Locations (1):
- University Medical Center, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valiev AG. [Features of secondary immune response and status of nonspecific resistance of the rat, fed rations with mare's milk, rich in essential fatty acids]. Vopr Pitan. 2001;70(5):10-3. Russian. PMID 11715690
- [Background] Pahud JJ, Mach JP. Equine secretory IgA and secretory component. Int Arch Allergy Appl Immunol. 1972;42(2):175-86. doi: 10.1159/000230604. No abstract available. PMID 4622991
- [Background] Foekel C, Schubert R, Kaatz M, Schmidt I, Bauer A, Hipler UC, Vogelsang H, Rabe K, Jahreis G. Dietetic effects of oral intervention with mare's milk on the Severity Scoring of Atopic Dermatitis, on faecal microbiota and on immunological parameters in patients with atopic dermatitis. Int J Food Sci Nutr. 2009;60 Suppl 7:41-52. doi: 10.1080/09637480802249082. Epub 2009 May 21. PMID 19462320
- [Background] Wulijideligen, Asahina T, Hara K, Arakawa K, Nakano H, Miyamoto T. Production of bacteriocin by Leuconostoc mesenteroides 406 isolated from Mongolian fermented mare's milk, airag. Anim Sci J. 2012 Oct;83(10):704-11. doi: 10.1111/j.1740-0929.2012.01010.x. Epub 2012 Mar 13. PMID 23035710
- [Background] Hancock JT, Salisbury V, Ovejero-Boglione MC, Cherry R, Hoare C, Eisenthal R, Harrison R. Antimicrobial properties of milk: dependence on presence of xanthine oxidase and nitrite. Antimicrob Agents Chemother. 2002 Oct;46(10):3308-10. doi: 10.1128/AAC.46.10.3308-3310.2002. PMID 12234868
- [Background] Palmer AC. Nutritionally mediated programming of the developing immune system. Adv Nutr. 2011 Sep;2(5):377-95. doi: 10.3945/an.111.000570. Epub 2011 Sep 6. PMID 22332080
- [Result] ADIYAR NURGAZIYEV, YERMEK AITENOV et al. Effect of mare's milk prebiotic supplementation on the gut microbiome and the immune system following antibiotic therapy // B IOD I V E R S I T A S.- Volume 21, Number 11, November 2020 Pages: 5065-5071 DOI: 10.13057/biodiv/d211110
- [Result] SAMAT KOZHAKHMETOV, DMITRIY BABENKO. The combination of mare's milk and grape polyphenol extract for treatment of dysbiosis induced by dextran sulfate sodium // B IOD I V E R S I T A S Volume 21, Number 5, May 2020 Pages: 2275-2280 DOI: 10.13057/biodiv/d210558
- [Result] Almagul Kushugulova, Samat Kozhakhmetov. Mare's milk as a prospective functional product //Functional Foods in Health and Disease. = 2018; 8(11): 537-543